CLINICAL TRIAL: NCT00406627
Title: Research for Elimination of Lymphatic Filariasis (ICIDR)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0137
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Lymphatic Filariasis
Keywords: filariasis, lymphatic filariasis, Egypt
MeSH Terms: conditions — Elephantiasis, Filarial; Filariasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to check blood samples for lymphatic filariasis to determine whether the recent Program to Eliminate Lymphatic Filariasis was successful in controlling lymphatic filariasis in areas of Egypt. Volunteers will participate in a health assessment program carried out by Ain Shams University and approved by the Egyptian Ministry of Health and Population. This program includes a brief interview and laboratory tests to detect worm parasites in participants' blood. Volunteers and family members found to have worms in their blood will be referred for treatment. This study will provide early detection of this parasitic infection and referral for prompt treatment in order to prevent spread of the infection to others. Approximately 23,500 people, 6 years of age and older, will participate per year. Study participants will include people living in areas of Egypt that are known to have the filariasis parasite. Volunteers will participate for up to 2 years.

DETAILED DESCRIPTION:
The purpose of this study is to detect lymphatic filariasis in blood samples to determine whether the recently concluded Program to Eliminate Lymphatic Filariasis has been successful in controlling lymphatic filariasis (LF) in areas of Egypt. The Research and Training Center on Vectors of Diseases (RTC) at Ain Shams University in Cairo, Egypt, will be the central site for data management and laboratory studies. Field sites (localities for village and school surveys) are 44 villages and small towns in 27 Districts and 7 governorates in the Nile river delta and in Giza. These localities are chosen based on inclusion in the Egyptian National Program to Eliminate Lymphatic Filariasis (PELF). Other localities will be chosen because of proximity to known endemic localities or a past history of filariasis endemicity. The primary study objective is to conduct population-based field studies to address key questions faced during late stages of programs for elimination of lymphatic filariasis (ELF). The investigators will test the hypothesis that filariasis has been eliminated in Egypt by 5 rounds of Mass Drug Administration (MDA) and attempt to answer the following questions: (1) Has LF been eliminated in localities included in the Egyptian National ELF Program? The investigators will study 44 localities (22 per year in alternate years). (2) What characteristics in endemic communities affect the likelihood of success or failure for ELF programs? The goal here is to identify key characteristics shared by localities that achieved elimination. (3) Are there significant foci of infection in localities that were not included in the Egyptian National PELF? The investigators will screen 20 new localities per year for the first 3 years of the project. The investigators will conduct a cohort study of the natural history of filarial antigenemia in treated populations. This study will test two hypotheses: (a) Filarial antigenemia without microfilaremia following completion of a MDA program with diethylcarbamazine and albendazole is of very little parasitological significance. That is to say, these people are unlikely to develop levels of microfilaremia that support filariasis transmission. (b) Following completion of a MDA program, filarial antigen levels in amicrofilaremic subjects will decline over time and disappear without further treatment. The investigators will assess the value of advanced diagnostic methods for detecting foci of continued transmission and for early detection of resurgent transmission. The duration of this study is 5 years, and approximately 23,500 people will participate per year. Most participants will be studied only once in cross-sectional surveys. The study population will include females and males over 6 years of age who live in areas of Egypt that are known to have been endemic or are now suspected to be endemic for bancroftian filariasis. Subject selection will not be based on health status. A subset of people, approximately 120, will be followed in a cohort study for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Gender, minority and child inclusion: Males and females will be included in population-based village studies without regard to race or ethnic group. There is no reason to exclude pregnant women from population-based studies. There is no reason to exclude children from the village/town studies, and they are included. Younger children will be studied in the school surveys (with large numbers per locality) because they are important sentinels for ongoing filariasis transmission.

Eligibility for the cohort study: Subjects in household surveys with positive immunochromotography test, filarial antigen tests, and negative microfilaria thick blood smears and who took diethylcarbamazine and albendazole during the Egyptian Program to Eliminate Lymphatic Filariasis will be invited to participate in the study. Subjects must be residents of localities that have met the Basic Elimination criterion (community microfilaria prevalence by thick smear less than 1% or antigen prevalence rate less than 2%). Consenting subjects will be screened further by testing a sample of venous blood collected after 9 p.m. for microfilaremia by membrane filtration and by performing an ELISA to quantitate filarial antigenemia in serum. Eligible subjects will have no microfilaremia by smear and antigen levels > 20 ng/ml.

Exclusion Criteria:

Exclusion of children less than 10 years of age from community studies of filarial antigen and microfilaria prevalence is justified because prevalence rates for these parameters are exceedingly low in young children in low transmission areas like Egypt.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117500
Dates: Start 2006-12; Study Completion 2011-12

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt